CLINICAL TRIAL: NCT00861679
Title: Therapy Protocol ALL SCT BFM International-open, Multicenter, Controlled, Prospective Study for Therapy and Therapy Optimisation in Patients With Acute Lymphoblastic Leukemia (ALL) and an Indication for Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Therapy Protocol Acute Lymphoblastic Leukemia Stem Cell Transplantation International
Acronym: ALL SCT BFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL-SCT-BFM-0321-08-HMO-CTIL
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2009-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: HSCT; ALL; GvHD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSCT from matched family or unrelated donors(MD) (Other): HSCT from matched family or unrelated donors(MD) to matched related donors.
  Interventions: Procedure: Transplantation with Stem Cells from Umbilical Cord

INTERVENTIONS:
Procedure: Transplantation with Stem Cells from Umbilical Cord — According to results from published experiences in children following suggestions are given:
  1. Number of Cells:
     * Number of nucleated cells infused exceed 2,5x10*7/kg recipient BW or
     * Number of nucleated cells collected exceed 3x10*7/kg BW
     * Number of CD34+ cells infused exceed 2x10*5/kg Recipient BW
  2. GVHD-prophylaxis:
     • MSD: CSA 3 mg/kg as described in the protocol + Prednisolone 1 mg/kg (day O to day 15, then tapering until day 28)
     • UD: as above + additional immunosuppression according to local protocols; ATG might increase risk of infectious complication and might be replaced by other drugs according to local protocols.
  3. HLA-matching for unrelated CB: a matched UB is defined by 6/6 HLA matches (A, B antigenic medium resolution and DRB1 allelic) and allocate to the transplantation group "MD". Less than 6/6 HLA matches allocate the patient to the "MMD" group.
  4. If many choices available ABO- major incompatibility should be avoided.

SUMMARY:
To evaluate whether HSCT from matched family or unrelated donors (MD) is equivalent to the HSCT from matched sibling donors (MSD). To evaluate the efficacy of HSCT from mismatched family or unrelated donors (MMD) as compared to HSCT from MSD/MD. To determine whether therapy has been carried out according to the main HSCT protocol recommendations. The standardisation of the treatment options during HSCT from different donor types aims at the achievement of an optimal comparison of survival after HSCT with survival after chemotherapy only. To prospectively evaluate and compare the incidence of acute and chronic GvHD after HSCT from MSD, from MD and from MMD.

ELIGIBILITY:
Inclusion Criteria:

all patients with ALL (except for patients with B-ALL) who fulfil the following criteria:

* age at time of initial diagnosis or relapse diagnosis, respectively

  ≤18 years
* indication for allogeneic HSCT
* complete remission (CR) is achieved before SCT
* written consent of the parents (legal guardian) and, if indicated, the minor patient via "Informed Consent Form"
* no pregnancy
* no secondary malignancy
* no previous HSCT
* HSCT is performed in a study participating centre.

Exclusion Criteria:

* not signed inform consent of the parents (legal guardian)
* pregnancy
* secondary malignancy
* previous HSCT

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 552 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
event-free and overall survival after allogeneic HSCT, occurrence of acute and chronic Graft-versus-Host-Disease (GvHD), occurrence and course of late effects after chemotherapy with subsequent allogeneic HSCT | 11 years

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center of Israel, Petach Tikvah, Israel